CLINICAL TRIAL: NCT02524457
Title: How Menopause Affects Lipid Metabolism in the Visceral Fat Depots
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD, phd-student, Rigshospitalet, Denmark
Other Study IDs: H-3-2014-096
Record Dates: First submitted 2015-08-11; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Insulin Sensitivity and Lipid Metabolism
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and fat biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Premenopausal: Premenopausal women going through gynecological surgery
  Interventions: Other: This is an observational study. There are no interventions
- Postmenopausal: Postemnopausal women going through gynecological surgery
  Interventions: Other: This is an observational study. There are no interventions
- Postmenopausal + HT: Postmenopausal women going through gynecological surgery who has been taking hormone treatment through the past year (as a minimum)
  Interventions: Other: This is an observational study. There are no interventions

INTERVENTIONS:
Other: This is an observational study. There are no interventions

SUMMARY:
The purpose of the study is to describe the molecular mechanisms related to an increased visceral fat mass and changed T-cell homeostasis. the project is expected to add new knowledge to the field of metabolic diseases after menopause and increase the focus of how lipid affects the development of metabolic disease in relation to the menopausal transition.

DETAILED DESCRIPTION:
The study is a cross sectional study including 60 women between 45 and 55 years of age. Investigators aim to include 20 premenopausal women, 20 postmenopausal women and 20 postmenopausal women taking hormone treatment (HT). All the women are going through gynecological surgery for benign reasons. During the operation investigators will take a visceral fat biopsy from the omentum.

maximally 1 month before- or after the operation the subject will meet at the lab for further testing, including:

* Health examination
* Blood samples
* OGTT
* DXA scan
* VO2 max testing
* MRI of the abdomen
* hyperinsulinemic euglycemic clamp

ELIGIBILITY:
Inclusion Criteria:

* women
* 45-55 years old
* for HT treated women (HT more than 1 year)

Exclusion Criteria:

* Infections during the last month
* chronic disease
* claustrophobia
* smoking
* Alcoholic intake > 14 servings
* hysterectomy before menopause
* oophorectomized
* early menopause (before 40 yrs)
* BMI > 30

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women from 45-55 years of age undergoing gynecological surgery for benign reasons.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 4 weeks
  measured through a hyperinsulinemic euglycemic clamp (Outcome: glucose infusion rate)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Abildgaard, MD, Principal Investigator — Rigshospitalet, Denmark

REFERENCES:
- [Background] Abildgaard J, Pedersen AT, Green CJ, Harder-Lauridsen NM, Solomon TP, Thomsen C, Juul A, Pedersen M, Pedersen JT, Mortensen OH, Pilegaard H, Pedersen BK, Lindegaard B. Menopause is associated with decreased whole body fat oxidation during exercise. Am J Physiol Endocrinol Metab. 2013 Jun 1;304(11):E1227-36. doi: 10.1152/ajpendo.00492.2012. Epub 2013 Apr 2. PMID 23548615
- [Background] Abildgaard J, Henstridge DC, Pedersen AT, Langley KG, Scheele C, Pedersen BK, Lindegaard B. In vitro palmitate treatment of myotubes from postmenopausal women leads to ceramide accumulation, inflammation and affected insulin signaling. PLoS One. 2014 Jul 7;9(7):e101555. doi: 10.1371/journal.pone.0101555. eCollection 2014. PMID 25000528